CLINICAL TRIAL: NCT02159261
Title: A Prospective Multicenter Non-interventional Study on Patients and Physicians Satisfaction of Yaz Plus
Brief Title: Assess Satisfaction of Patients and Physicians With Results of Yaz Plus Treatment for 13 Cycles
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17177; YZ1410RU (Other: Company Internal)
Record Dates: First submitted 2014-06-06; First posted 2014-06-09 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Contraception
Keywords: Personal Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Female patients ≥ 18 years old requiring contraception.
  Interventions: Drug: BAY98-7071_EE20/DRSP/L-5-MTHF

INTERVENTIONS:
Drug: BAY98-7071_EE20/DRSP/L-5-MTHF — Patients treated by Physicians under approved local prescriptions

SUMMARY:
Local prospective multicenter non-comparative non-interventional observational study. It's planed to assess satisfaction of patients and physicians with results of Yaz Plus treatment for 13 cycles in real practice.

DETAILED DESCRIPTION:
Non-interventional, Yaz Plus, Contraception, Assess satisfaction, Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥ 18 years old
* Requiring contraception
* Prescribed with Yaz Plus for the first time

Exclusion Criteria:

* Contraindications for the use of Yaz Plus in accordance with the local product information

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients ≥ 18 years old requiring contraception, treated with Yaz Plus for the first time and for which the inclusion and exclusion criteria are fulfilled, are eligible for enrolment into the study.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2014-07-15 (Actual); Primary Completion 2016-08-14 (Actual); Study Completion 2016-08-14 (Actual)

PRIMARY OUTCOMES:
Satisfaction measured with a Likert response scale (from 1 - poor to 5 - excellent) | Up to 12 months

SECONDARY OUTCOMES:
Changes in EVAPIL scale for assessment of tolerability of oral contraceptives. | Baseline to 12 months
Number of participants with adverse events as a measure of safety and tolerability | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Russia